CLINICAL TRIAL: NCT05772780
Title: The Effect of Varied MP-3 Biofeedback Training on Visual Functions in Central Vision Loss: a Randomized Trial
Brief Title: MP-3 Biofeedback Training and Central Vision Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amore Filippo (Other)
Responsible Party: Sponsor-Investigator, Amore Filippo, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4172
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Training will be performed for two days a week
  Interventions: Device: MP-3 microperimeter
- Group B (Experimental): Training will be performed three days a week
  Interventions: Device: MP-3 microperimeter

INTERVENTIONS:
Device: MP-3 microperimeter — Biofeedback stimulation two days a week
Device: MP-3 microperimeter — Biofeedback stimulation three days a week

SUMMARY:
The objectives of this investigation are:

* evaluate the results of rehabilitation treatment using photostimulation with a structured stimulus in two different samples of low vision subjects with central vision loss who will be subjected to biofeedback at the MP3 microperimeter with different timing;
* compare the effectiveness of the rehabilitation treatments in the two groups to provide useful indications for proposing standardisation of the rehabilitation pathway focusing on photostimulation in subjects with central vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Age related macular degeneration

Exclusion Criteria:

* Cognitive impairment; concomitant eye disease; significant media opacities; ocular surgery within previous 90 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Fixation stability | 6 months
  Achievement of a stable fixation, defined according to Fuji classification (Stable: if more than 75% of the fixation points are inside a 2° diameter circle that has as a center the centroid of all fixation points) and the Bivariate Contour Ellipse Area, were selected as primary outcomes.
Reading speed | 6 months
  Achievement of good reading speed: higher than 87 words per minutes was defined as our secondary outcome. Parameters for words per minutes are referred to visually impaired functional reading reported in literature

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No